CLINICAL TRIAL: NCT06470945
Title: Clinical Assessment of the Color Stability of Sectional and Full Glass Ceramic Laminate Veneer by Using Digital Shade Matching Device. A Randomized Clinical Trial
Brief Title: Color Stability of Sectional and Full Glass Ceramic Laminate Veneer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Aya mahmoud, Dr., October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Spacing of Anterior Teeth
Keywords: porcelain fragments; miniveneers; sectional veneers; laminate veneers; partial veneers

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data analyst and statistician will be blinded and The patient will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention- Glass ceramic sectional veneer (Experimental): participants receive Glass ceramic sectional veneer covering only the area of defect
  Interventions: Procedure: Glass ceramic sectional veneer
- control- Glass ceramic laminate veneer (Active Comparator): participants receive laminate veneers made of glass ceramics as a gold standard
  Interventions: Procedure: Glass ceramic laminate veneer

INTERVENTIONS:
Procedure: Glass ceramic sectional veneer — partial laminate veneer
  Arms: intervention- Glass ceramic sectional veneer
Procedure: Glass ceramic laminate veneer — Glass ceramic laminate veneer
  Arms: control- Glass ceramic laminate veneer

SUMMARY:
The aim of the study is to evaluate the color stability of full and sectional glass ceramic laminate veneer as esthetic failure is reported to be common failure in laminate following clinical service.

The null hypothesis is that there will be no apparent change in color stability between full and sectional veneer over one year of clinical service

DETAILED DESCRIPTION:
The success of any esthetic restorative material depends primarily on the color match and then on the color stability of the material. color changes by time reduce the longevity and quality of restorations.

This in vivo study planned to evaluate the color stability of full and sectional glass ceramic laminate veneer using a digital shade device The primary objective of the study to evaluate the color stability of sectional glass ceramic veneer compared to full laminate veneer

ELIGIBILITY:
Inclusion Criteria:

Patients seeking for esthetics with the following criteria:

1. Male or female patients age range above 18 years old
2. Minor esthetic defects in anterior region
3. Multiple spacing, diastemas
4. Incisal fracture
5. Initial proximal caries
6. Patients able physically and psychologically to tolerate restorative procedures
7. Patients willing to return for follow-up examinations and evaluation
8. Class I occlusion

Exclusion Criteria:

* Patients free of

  1. Tempromandibular disorders
  2. Para-functional habits
  3. Cracked teeth
  4. Moderate or deep caries
  5. Heavily discolored teeth
  6. Heavy smokers
  7. Enamel defects compromising bonding
  8. Active periodontal disease
  9. Pulpal disease
  10. Mobility
  11. Occlusal disturbances
  12. Class II and III occlusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Color change | Baseline,3,6,9,12 months
  assessment of color change using spectrophotometer

SECONDARY OUTCOMES:
shade match | Baseline,3,6,9,12 months
  assessment of shade match using Modified USPHS

CONTACTS AND LOCATIONS:
Overall Officials: Aya M Ali, BDS, Principal Investigator — October University for Modern Sciences & Arts
Locations (1):
- October University for Modern Sciences & Arts, Giza, Giza,6th October City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided